CLINICAL TRIAL: NCT02093585
Title: Changes in Coagulation and Platelet Reactivity in HIV-1 Infected Patients Switching Between Abacavir and Tenofovir Containing Antiretroviral Regimens
Brief Title: Tenofovir Abacavir Platelet Activation Study
Acronym: TAPAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jan Gerstoft (Other)
Responsible Party: Sponsor-Investigator, Jan Gerstoft, MD, DMSc, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2013-001685-42
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: HIV
Keywords: HIV-1; Abacavir; Platelet activation; Thromboelastography; Coagulation
MeSH Terms: conditions — Thrombosis | interventions — abacavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir to abacavir (Experimental): Patients switching from tenofovir (245 mg QD) to abacavir (600 mg QD)
  Interventions: Drug: abacavir (600 mg QD)
- Abacavir to tenofovir (Experimental): Patients switching from abacavir (600 mg QD) to tenofovir (245 mg QD)
  Interventions: Drug: tenofovir (245 mg QD)

INTERVENTIONS:
Drug: abacavir (600 mg QD)
  Arms: Tenofovir to abacavir
Drug: tenofovir (245 mg QD)
  Arms: Abacavir to tenofovir

SUMMARY:
Some but not all observational studies have found that current exposure to abacavir is associated with increased risk of cardiovascular events such as myocardial infarction, stroke and cardiovascular death. This study aim to investigate possible adverse effect of abacavir on platelet reactivity, coagulation and endothelial activation in HIV-1 infected patients. The study is an open-labeled cross-over trial, where patients receiving antiretroviral therapy containing abacavir switch treatment to a regimen containing tenofovir and vice versa for a period of 90 days.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Can understand and sign written informed consent
* Received one of the above mentioned antiretroviral regimens continuously ≥ 6 months
* HIV RNA < 400 copies/mL for ≥ 6 months

Exclusion Criteria:

* Receiving anticoagulant therapy, adenosine diphosphate (ADP) receptor inhibitors, aspirin or nonsteroidal antiinflammatory drugs (NSAIDs)
* Previous ischemic heart disease, peripheral atherosclerotic disease or stroke
* Coagulation disorder (e.g. hemophilia, factor V Leiden mutation)
* Platelet count < 150 x 109/L during the past 6 months from inclusion
* Estimated glomerular filtration rate (eGFR) <70 during the past 6 months from inclusion
* Humane leukocyte antigen (HLA)-B*57:01 positive genotype
* Hepatitis B or C positive during the past year from inclusion
* Hypersensitivity to the active substances or to any of the excipients

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Differences in platelet aggregation (Multiplate) before and after switching between abacavir and tenofovir. | before and after 90 days intervention
Differences in clot formation kinetics (thromboelastography) before and after switching between abacavir and tenofovir. | before and after 90 days intervention

SECONDARY OUTCOMES:
Concentration of plasma lipids | Before and after 90 days intervention
activated partial thromboplastin time (APTT) | 90 days
international normalized ratio (INR)/Factor II, VII, X | Before and after 90 days intervention
Platelet count | Before and after 90 days intervention
Fibrinogen | Before and after 90 days intervention
D-dimer | Before and after 90 days intervention
Antithrombine | Before and after 90 days intervention
Interleukin 6 (IL-6) | Before and after 90 days intervention
High sensitivity C reactive protein (HS-CRP) | Before and after 90 days intervention
Soluble P-Selectin | Before and after 90 days intervention
soluble CD40 ligand (sCD40L) | Before and after 90 days intervention
Syndecan-1 | Before and after 90 days intervention
Soluble E-selectin | Before and after 90 days intervention
Tissue plasminogen activator | Before and after 90 days intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gerstoft, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Klinik for Infektionsmedicin og Reumatologi, 8622, Copenhagen Ø, Copenhagen, Denmark